CLINICAL TRIAL: NCT01482182
Title: Prediction of Chemotherapy Response and Patient Prognosis in Non-small Cell Lung Cancer: Dynamic Contrast-enhanced MRI and Diffusion-weighted Imaging Versus Volume-based Parameter of 18F-FDG PET
Brief Title: Predictive Value of FDG PET/CT, DWI and DCE-MRI Scans for Non-small Cell Lung Cancer Patients Receiving Chemotherapy
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-05-087
Record Dates: First submitted 2011-11-17; First posted 2011-11-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Diffusion-weighted MRI; 18F-FDG PET; Treatment response; Prognosis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this prospective study, the investigators will evaluate and compare the usefulness of functional and volumetric informations obtained by 18F-FDG PET and MRI before and after the palliative chemotherapy with the aim of predicting tumor response and prognosis in patients with advanced Non-small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Study cohort will undergo PET/CT and MRI scans prior to chemotherapy and after the first chemotherapy cycle. MRI scans include DCE-MRI and DWI. The following parameters will be calculated using these values:

1. Metabolic parameters on FDG-PET A. SUV change ratio (SCR) = SUVpost/SUVpre B. MTV change ratio (VCR) = MTVpost/pre C. TLG change ratio = SCR X VCR
2. Perfusion parameters on DCE-MRI A. Kep B. K-trans C. ve
3. Diffusion parameters on DWI A. Mean ADC B. fDM

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NSCLC
* Newly diagnosed Stage stage IV
* Participant is being considered for the chemotherapy with EGFR TKI as a first line therapy
* At least one measurable primary or other intrathoracic lesion >= 2cm, according to RECIST
* Performance status of 0 to 2 on the ECOG scale
* Age 18 years or older
* Able to tolerable PET/CT and MRI imaging required by protocol
* Able to give study-specific informed consent

Exclusion Criteria:

* Pure bronchioloalveolar cell carcinoma histology
* Thoracic radiotherapy, lung surgery or chemotherapy within three months prior to inclusion in the study
* Poorly controlled diabetes
* Prior malignancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
DWI, DCE-MRI, and FDG PET as early predictor for response and prognosis | one year
  The primary endpoint of this study is the prediction of one-year overall survival by monitoring the metabolic and functional responses of the tumor following one cycle of chemotherapy.

SECONDARY OUTCOMES:
Correlation among DWI, DCE-MRI, and FDG PET and relationship with prognosis | one year
  Correlation among metabolic response, functional response on MRI, and standard anatomic response using the RECIST criteria
Correlation among DWI, DCE-MRI, and FDG PET and relationship with prognosis | one year
  (i) the correlation among metabolic response, functional response on MRI, and standard anatomic response using the RECIST criteria (ii) the correlation between functional response (metabolic and MR parameters) and progression-free survival (iii) comparison between the predictive values of FDG-PET and MRI for one-year overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Yun Lee, Dr., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea